CLINICAL TRIAL: NCT06668896
Title: An Open-Label, Four-Treatment, Parallel Study of the Comparative Pharmacokinetics of a Progesterone Intravaginal Ring (IVR) 8 mg and 12 mg/Day Versus Progesterone Vaginal Insert 100mg
Brief Title: Comparing the Pharmacokinetics of a Progesterone Ring Versus a Progesterone Vaginal Insert
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DARE-PTB1-001; 1R44HD101169-01A1 (NIH)
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pre Term Birth
Keywords: normal healthy
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DARE-PTB1 8mg IVR (Experimental): Intravaginal ring containing 8mg progesterone administered once for 14 days.
  Interventions: Drug: Progesterone
- DARE-PTB1 12mg IVR (Experimental): Intravaginal ring containing 12mg progesterone administered once for 14 days.
  Interventions: Drug: Progesterone
- DARE-PTB1 12mg IVR every 3 days (Experimental): Intravaginal ring containing 12mg progesterone administered every 3 days for 15 days.
  Interventions: Drug: Progesterone
- Endometrin 100mg (Active Comparator): 100mg progesterone vaginal insert, three times daily for 14 days.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Each arm will administer different amounts of progesterone vaginally (8mg to 100mg) over a 14-15 day time period.

SUMMARY:
This study is looking for healthy female adults to use an vaginal ring with differing amounts of the hormone progesterone and go through a series of blood draws to measure how much progesterone is in the body following the use of these vaginal rings over an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Individuals assigned female at birth who are post-menopausal, women 40 to 65 years of age, inclusive. Postmenopausal is defined as 6-months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL (if not taking systemic hormone therapy) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Able and willing to correctly and independently complete all study procedures.
* Able to read, understand, and provide written informed consent after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures.
* VA vaginal pH of ≤ 5.0. Women with vaginal atrophy may rescreen at least 6 weeks after starting either systemic or topical estradiol therapy.
* Women who are taking systemic (e.g. oral, injectable, transdermal) progesterone (P4) therapy must have at least 2 weeks of wash out from the last dose prior to visit 2.

Exclusion Criteria:

* Subjects with clinically significant chronic kidney disease defined as Glomerular Filtration Rate of <60 mL/min/1.73m2
* Subjects with uninvestigated hematuria
* Subjects with known nephrolithiasis, known polycystic kidney disease (PKD), or other known renal genetic disorders
* Subjects with prior pelvic malignancies requiring radiation therapy, or whose surgery for such has led to complications such as fistulas, etc.
* Subjects with a history of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or study treatment administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial. This includes but is not limited to the following:

  * Active chronic hepatitis B or hepatitis C infection including hepatitis B surface antigen and hepatitis C antigen positive patients with or without abnormal liver enzymes
  * Concurrent neurodegenerative disease
  * Cardiovascular: uncontrolled hypertension, unstable angina, myocardial infarction or symptomatic congestive heart failure within the past 6 months or serious uncontrolled cardiac arrhythmia or use of Class 1 antiarrhythmic
  * Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol
* Subjects with hypersensitivity toward any ingredients in the study treatments.
* Participation in any other investigational drug or device trial in which administration of an investigational study drug/device occurred within 30 days or placement of a non-drug eluting medical device within 15 days prior to the Screening Visit (Visit 1). This does not include re-enrollments into this study, who require at least 14 days of washout prior to re-enrollment.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Systemic pharmacokinetics of progesterone, Concentration over 24 hours | 14 days
  Describe the concentration of progesterone (P4) in blood prior to, during and after 24 hours of DARE-PTB1 IVR (8mg and 12mg) over 14 days of use.